CLINICAL TRIAL: NCT05727813
Title: Early Breast Cancer Ultrasound-guided Visual-ICE Galil Cryoablation; Can Tumor Cell Death Induced by Cryoablation be Detected by Specific Circulating Markers?
Brief Title: To Detect Cryoimmunologic Response Induced by Early Breast Cancer Ultrasound-guided Cryoablation (ICE-study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, federica pediconi, Prof. Federica Pediconi, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URomLS Prot.0930/2021Rif. 6528
Record Dates: First submitted 2023-01-03; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cancer, Treatment-Related; Tumor of Breast; Systemic Inflammatory Response; Stage I Breast Cancer
Keywords: breast cancer treatment; Breast imaging evaluation; immunologic response; cryotherapy
MeSH Terms: conditions — Neoplasms, Second Primary; Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryoablation (Experimental): We will enroll women with a biopsy-proven diagnosis of early-stage breast cancer (T1 N0), not eligible for neo-adjuvant therapy, scheduled to breast surgery (mastectomy or nodulectomy), who have given the informed consent for the study.
  We will recruit 20 women who will undergo cryoablation.
  Interventions: Device: cryoablation
- no cryoablation (No Intervention): The results will be compared with those obtained from a control group of 20 women, who will follow the same therapeutic pathway for the treatment of breast cancer without performing cryoablation.

INTERVENTIONS:
Device: cryoablation — cryoablation of breast cancer smaller than 2 cm
  Arms: cryoablation

SUMMARY:
The aim of our study is to examine the cryoimmunologic response and its mechanisms induced by US-guided cryoablation of small breast tumors (<2 cm) not eligible to neoadjuvant therapy. We will recruit 30 women who will undergo cryoablation and their results will be compared with a control group of 30 women, who will follow the same therapeutic pathway without performing cryoablation. All recruited patients will undergo an enrollment check, pre-cryoablation breast MRI and blood test to assess immune response, breast cancer US-guided cryoablation, post-cryoablation breast MRI and the same blood test to evaluate immunologic response. Within 21 days all patients will undergo breast surgery, with immuno-histopathological analysis on surgical specimen.

At least 10 days after surgery the patient will undergo clinical breast examination, blood test to assess immune response and patient satisfaction questionnaire.

Cryoablation treatment will be performed using a 14G cryoprobe under us-guidance for visualization of the ice ball surrounding the lesion. The ultrasound guide is used to ensure that the action affects the entire tumor and that therapeutic temperatures are reached in every part of the tumor.

Pre- and post- cryoablation breast MRI will be performed on a 3T magnet to assess cryoablation rate of success. Artificial intelligence algorithms will also be used for this purpose. Cryoablation treatment efficacy will also be evaluated with ultrasound.

The immunological fitness of cancer patients will be studied by flow cytometry, evaluating the presence of cytokines/chemokines relevant during anticancer immune response/tumor progression and for the presence of molecules released by cells during an immunogenic cell death.

The goal of our study will be to demonstrate that cryoablation of breast cancer can induce an antitumor immune response.

Therefore this approach could become an additional tool in the oncological treatment of breast cancer.

DETAILED DESCRIPTION:
We will enroll women with a biopsy-proven diagnosis of early-stage breast cancer (T1 N0), not eligible for neo-adjuvant therapy, scheduled to breast surgery (mastectomy or nodulectomy), who have given informed consent for the study.

We will recruit 30 women who will undergo cryoablation. Their results will be compared with those obtained from a control group of 30 women, who will follow the same therapeutic pathway for the treatment of breast cancer without performing cryoablation.

The primary objective of our study is the characterization of the Immunogenic Cell Death (ICD) induced, the inflammatory response and the modulation of circulating T immune cells induced by tumor cryoablation treatment in the serum of breast cancer patients.

The circulating ICD biomarkers HMGB1, calreticulin and HSP70/90 will be analysed and also the profile of Th1 and Th2 type cytokines (IFN-γ, IL-12 (p40/p70), IL-15, IL-17, IL-2, IL-7, IP-10, IL-13, IL-5, IL-4), pro-inflammatory cytokines (IL-1α, IL-1β, IL- 6, TNF-α, IL-1RA, IL-2R, IL-8, CRP, IL-17, IFN-α), immunosuppressive cytokines (TGF-β1, IL-10, PGE2), chemokines (CCL5/RANTES, CCL3/MIP-1α, CCL4/MIP-1β, CCL2/MCP-1, CXCL9/MIG, CCL11/Eotaxin). Immune cell subsets will be characterized by flow cytometry: besides the conventional immune cell subsets (NK, Monocyte, Granulocyte, T and B cells), specific T cell subsets (Treg, naïve, memory, central effector) will be characterized and also the expression of immune markers associated to activation (CD137) or suppression/exhaustion (PD1, CTLA4, TIM3, LAG3).

Secondary endpoints are:

1. Cryoablation treatment efficacy and safety

   We will evaluate Recist criteria rate of complete response to cryoablation with breast ultrasound and breast MRI. Incidence vand severity of complications related to cryoablation will be monitored to establish safety profile ablating breast cancer with 10 mm margins around the primary tumor.
2. Cryoablation treatment capability to induce immunogenic tumor cell death.

   The presence and the extent of tumor necrosis / apoptosis on surgical specimen sections stained with hematoxylin-eosin will be evaluated. Immunohistochemical tests will be used to verify the activation of apoptotic mechanisms and Immunogenic cell death activation.
3. Tumor microvesicles release following Cryoablation treatment. During cell death, microvesicles (MVs) released by the cell transport a complex molecular cargo that can act as source of antigen repertoire and activatory signals to Antigen Presenting cells (APCs). Tumor derived MVs released in the serum of the patients will be isolated by ultracentrifugation steps as preliously described. The isolated MVs will be tested for the expression of Calreticulin and HMGB1.

All enrolled patients will undergo series of check as shown below (ICE-STUDY STEPS) :

enrollment check (STEP 0), breast MRI pre-cryoablation treatment (STEP 1) and post-cryoablation treatment (STEP 4), breast cancer US-guided cryoablation

(STEP 2), blood test to assess immune response (STEP 1, STEP 3, STEP 4, SURGERY and STEP 5) and surgical specimen immuno-histopathological analysis.

Enrollment check (STEP 0) will be conducted by a radiologist and an oncologist, where the patient's medical history will be collected and a breast examination of the affected site will be performed. The patient will also undergo breast US to evaluate cryoablation treatment feasibility (distance >1 cm between the tumor and the skin, the nipple or the chest wall). If the patient is considered eligible to the study, the protocol will be illustrated in detail and informed consent will be collected.

Breast MRI will be performed pre-cryoablation (STEP 1) and post-cryoablation (STEP 4) to assess Visual-ICE ablation rate of success. Artificial intelligence algorithms will also be used for this purpose. Cryoablation treatment efficacy will also beevaluated with ultrasound (STEP 4).

STEP 2 consists in US-guided cryoablation treatment of the breast lesion.

Within 21 days from the enrollment the patient will undergo breast surgery and blood test.

During the Final STEP, the patient will undergo clinical breast examination, blood test to assess immune response and patient satisfaction questionnaire.

ICE-STUDY STEPS:

STEP 0: enrollment check

* Imaging: US
* Assessment:

  1. consent
  2. breast biopsy with histological result
  3. clinical history
  4. laboratory results
  5. clinical breast examination
  6. pharmacological therapy

STEP 1: Within 10 days from STEP 0

* Imaging: MRI (pre-cryoablation treatment)
* Assessment:

  1. blood test for immune response
  2. side effects

     STEP 2: CRYOABLATION (At least 24h after MRI)
* Assessment:

  1. cryoablation complications and side effects

     STEP 3: Blood test for immune response (48/72 h after cryoablation)

STEP 4: After 7 days from cryoablation and before surgery

* Imaging: MRI and/or US (post-cryoablation treatment)
* Assessment:

  1. patient satisfaction questionnaire.
  2. Side effects
  3. pharmacological therapy
  4. clinical breast examination
  5. blood test for immune response

SURGERY: Within 21 days from STEP 0

* Assessment:

  1. surgery
  2. complications
  3. specimen histological evaluation
  4. blood test for immune response

     STEP 5 - FINAL: At least 10 days after surgery
* Assessment:

  1. patient satisfaction questionnaire
  2. side effects
  3. pharmacological therapy
  4. clinical breast examination
  5. blood test for immune response

All cryoablation sessions will be performed under US-guidance by a single board-certi¿ed interventional radiologist. Biopsy, percutaneous cryoablation will be carried out using an argon-based cryoablation unit (BTG Cryoablation System).

Both preoperative US and MRI images will be compared in order to determine the correct positioning of the probe for tumor ablation. All the procedures will be carried out under local anesthesia given by injection of 2-5mL of 2% lidocaine proximal to the tumor lesion and along the course of the cryoprobes. One or more cryoprobes will be inserted into the targeted tumor using US guidance, through a small skin incision of 1-2mm. To avoid cryoinduced skin injury and facilitate the ablation of breast tissue at least 1cm beyond all apparent tumor margins, warming bags will be placed on the breast skin.

Due the relatively low heat load of breast parenchyma compared with internal organs, it was estimated that 1cm of visible ice beyond all the tumor margins would be necessary to generate cytotoxic temperatures (e.g.,-40¿C) throughout the breast tumor.

Each cryoablation treatment session consists in two cycles of 8 minutes of duration, followed by a 4-minute active thawing phase and a 4-minute passive thawing phase. The latter is considered useful to maximize cell death. US guidance will be also used to verify the formation of a homogeneous hypoechoic area, owing to the iceball, which encompassed the tumor all around and to detect early complications. The probes will be removed after the second phase of thawing, without the need for skin suture. After the procedure, the patients will be discharged in 2 hours a¿er the ablation, without any prescription.

The clinical outcome will be evaluated with US at the end of the cryoablation procedure and 7 days a¿er with clinical examination and MRI. The absence of such signs or symptoms will be interpreted as an optimal clinical result.

Immunogenic CELL DEATH and Inflammatory circulating Biomarkers will be analysed at different time points (5 time points:

before, 48 h and 7 days after cryoablation; before and after 10 days from surgery). Plasma will be isolated by EDTA treated blood (10 ml/sample) by centrifugation (4000 rmp/5'/4°C) and aliquoted and stored at -80°C.

The ICD biomarkers characterized will be: calreticulin, HMGB1, HSP70/90 (by ELISA and/or chemioluminescence immune sandwich tests).

Circulating Inflammatory mediators will also be analyzed by xMAP Multiplex platform including the following molecules:

Th1 and Th2 type cytokines (IFN-γ, IL-12 (p40/p70), IL-15, IL-17, IL-2, IL-7, IP-10, IL-13, IL-5, IL-4), pro-inflammatory

cytokines (IL-1α, IL-1β, IL-6, TNF-α, IL-1RA, IL-2R, IL-8, CRP, IL-17, IFN-α), immunosuppressive cytokines (TGF-β1, IL- 10, PGE2), chemokines (CCL5/RANTES, CCL3/MIP-1α, CCL4/MIP-1β, CCL2/MCP-1, CXCL9/MIG, CCL11/Eotaxin)] will be analyzed.

The samples of each patient will be analysed for each biomarker simultaneously to avoid inter-experiment bias.

Microvesicles will be isolated by ultracentrifugation steps in micro-method scale (2 mL of plasma) and the analysis of calreticulin and HMGB1 will be performed by flow cytometry/ELISA (3 Time point: before, 48h and at the end of the procedure) Immune phenotyping will be performed by mulitparametric flow cytometry, characterizing the immune cell subsets(NK, T, B cells, granulocyte, monocytes). T cell subsets will be specifically characterized for Treg (CD25/foxp3), Naive/memory effector memory T cell (CCR7/CD45RA) and for activatory or exhausted phenotype (CD137, ICOS, PD1, CTLA4, TIM3, LAG3).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 year-old women with needle (14-20 G) biopsy-proven invasive breast cancer. The specimens taken are adequate for tumor classification and receptors analysis;
* imaging (ultrasound and magnetic resonance imaging) confirmed single <2 cm breast cancer;
* clearly visible lesion on ultrasound with a minimum distance of 1 cm between the tumor and the skin and 2 cm between the tumor and the nipple;
* not eligible patients for neo-adjuvant therapy;
* patients who are scheduled for breast cancer surgical resection (lumpectomy or mastectomy) after cryoablation; stage I disease: T1 N0;

Exclusion Criteria:

* DCIS without invasive components on the core biopsy;
* Tamoxifen, aromatase inhibitors and neoadjuvant chemotherapy within 30 days prior to Visual-ICE treatment;
* XRT or previous ablative therapy to the affected breast;
* distance <1 cm between the tumor and the skin, the nipple or the chest wall;
* microcalcifications as the only evidence of breast cancer on imaging;
* breast implants;
* severe cardiac or cerebrovascular disease;
* pregnancy, nursing or puerperium;
* patients with a general health status ASA> 2, which includes in a non-limiting way patients suffering from renal dysfunction due to hepatorenal syndrome or who are in the perioperative period for liver transplantation;
* active and ongoing infection, e.g. urinary tract infection, respiratory tract infection and other known infections;
* poor blood glucose control;
* severe hypertension;
* any contraindications for Visual-ICE ablation therapy;
* sleep apnea syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer patients
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Immunogenic Cell Death induced by tumor cryoablation, cytokines | 12 months
  Characterization of the Immunogenic Cell Death induced by tumor cryoablation treatment in the serum of breast cancer patients.
  Evaluation of serum modifications of the following molecules:
  Th1 and Th2 type cytokines (IFN-γ, IL-12 (p40/p70), IL-15, IL-17, IL-2, IL-7, IP-10, IL-13, IL-5, IL-4)
Immunogenic Cell Death induced by tumor cryoablation, pro-inflammatory cytokines | 12 months
  Characterization of the Immunogenic Cell Death induced by tumor cryoablation treatment in the serum of breast cancer patients.
  Evaluation of serum modifications of the following molecules:
  pro-inflammatory cytokines (IL-1α, IL-1β, IL-6, TNF-α, IL-1RA, IL-2R, IL-8, CRP, IL-17, IFN-α),
Immunogenic Cell Death induced by tumor cryoablation, immunosuppressive cytokines | 12 months
  Characterization of the Immunogenic Cell Death induced by tumor cryoablation treatment in the serum of breast cancer patients.
  Evaluation of serum modifications of the following molecules:
  immunosuppressive cytokines (TGF-β1, IL-10, PGE2),
Immunogenic Cell Death induced by tumor cryoablation, chemokines | 12 months
  Characterization of the Immunogenic Cell Death induced by tumor cryoablation treatment in the serum of breast cancer patients.
  Evaluation of serum modifications of the following molecules:
  chemokines (CCL5/RANTES, CCL3/MIP-1α, CCL4/MIP-1β, CCL2/MCP-1, CXCL9/MIG, CCL11/Eotaxin),
Immunogenic Cell Death induced by tumor cryoablation, ATP and HMGB1 | 12 months
  Characterization of the Immunogenic Cell Death induced by tumor cryoablation treatment in the serum of breast cancer patients.
  Evaluation of serum modifications of the following molecules: ATP and HMGB1 are molecules released in the serum by cancer cells during immunogenic cell death.

SECONDARY OUTCOMES:
Rate of complete response | 12 months
  Evaluate Recist criteria rate of complete response to cryoablation with breast ultrasound and breast MRI
Cryoablation treatment capability to induce immunogenic tumor cell death, specimen | 12 months
  Analyzing surgical specimen sections stained with hematoxylin-eosin, the presence and the extent of tumor (cm) necrosis will be evaluated.
safety margin of Cryoablation treatment | 12 months
  ablating breast cancer with 5-10 mm margins around the primary tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Pediconi, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sabel MS, Nehs MA, Su G, Lowler KP, Ferrara JL, Chang AE. Immunologic response to cryoablation of breast cancer. Breast Cancer Res Treat. 2005 Mar;90(1):97-104. doi: 10.1007/s10549-004-3289-1. PMID 15770533
- [Result] Mauri G, Sconfienza LM, Pescatori LC, Fedeli MP, Ali M, Di Leo G, Sardanelli F. Technical success, technique efficacy and complications of minimally-invasive imaging-guided percutaneous ablation procedures of breast cancer: A systematic review and meta-analysis. Eur Radiol. 2017 Aug;27(8):3199-3210. doi: 10.1007/s00330-016-4668-9. Epub 2017 Jan 3. PMID 28050693
- [Result] McArthur HL, Diab A, Page DB, Yuan J, Solomon SB, Sacchini V, Comstock C, Durack JC, Maybody M, Sung J, Ginsberg A, Wong P, Barlas A, Dong Z, Zhao C, Blum B, Patil S, Neville D, Comen EA, Morris EA, Kotin A, Brogi E, Wen YH, Morrow M, Lacouture ME, Sharma P, Allison JP, Hudis CA, Wolchok JD, Norton L. A Pilot Study of Preoperative Single-Dose Ipilimumab and/or Cryoablation in Women with Early-Stage Breast Cancer with Comprehensive Immune Profiling. Clin Cancer Res. 2016 Dec 1;22(23):5729-5737. doi: 10.1158/1078-0432.CCR-16-0190. Epub 2016 Aug 26. PMID 27566765
- [Derived] Galati F, Pasculli M, Maroncelli R, Rizzo V, Moffa G, Cerbelli B, d'Amati G, Catalano C, Pediconi F. Ultrasound-guided cryoablation of early breast cancer: safety, technical efficacy, patients' satisfaction, and outcome prediction with MRI/CEM: a pilot case-control study. Eur Radiol Exp. 2024 Oct 22;8(1):120. doi: 10.1186/s41747-024-00515-4. PMID 39436590